CLINICAL TRIAL: NCT05517395
Title: The Effectiveness of Health Belief Model Based Education Program on Improve Knowledge and Behaviors Related to Undernutrition Among Mothers With Children Under Two Years in Indonesia
Brief Title: The Effectiveness of HBM-based Education Program on Improve Knowledge and Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, Ph.D, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202208020
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Undernutrition; Stunting; Wasting; Underweight
Keywords: Undernutrition; Health belief model; Children
MeSH Terms: conditions — Malnutrition; Growth Disorders; Cachexia; Thinness

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial design with one intervention arm (nutrition education and complementary feeding) and one control (usual care) arm (1:1 ratio).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization will be performed by a research assistant with no access to participant information and who did not participate in the enrolment process. The person performing the intervention will be blinded to group allocation. Outcome data will be collected by another two blinded research assistants, one for the intervention group and one for the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health nutrition education (Experimental): The participants in intervention group will receive health nutrition education based on a health belief model including nutrition health education (booklet), and telephone call support.
  Interventions: Behavioral: health nutrition education
- usual care (Active Comparator): Control group will only receive usual care. Usual care is routine measurement of children including height, length, weight, head circumference, monitoring children's activities, and monitoring the immunization status of children.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: health nutrition education — The participants in intervention group will receive health nutrition education based on a health belief model including nutrition health education (booklet), and telephone call support.
  Arms: health nutrition education
Behavioral: usual care — Control group will only receive usual care. Usual care is routine measurement of children including height, length, weight, head circumference, monitoring children's activities, and monitoring the immunization status of children.
  Arms: usual care

SUMMARY:
The randomized controlled trial design with one intervention arm (nutrition education and complementary feeding) and one control (usual care) arm (1:1 ratio). Randomization of each participant to the groups will be carried out using Random Allocation Software 1.0 (https://random-allocation-oftware.software.informer.com/1.0/) to intervention or control groups in a 1:1 ratio. The sample size to be recruited is 80 participants.

DETAILED DESCRIPTION:
The randomized controlled trial design with one intervention arm (nutrition education and complementary feeding) and one control (usual care) arm (1:1 ratio). will be conducted in the second phase. This trial will be conduct in mothers with children aged under 2 years of age of Nusa Tenggara Barat Province of Indonesia.

Randomization of each participant to the groups will be carried out using Random Allocation Software 1.0 (https://random-allocation-oftware.software.informer.com/1.0/) to intervention or control groups in a 1:1 ratio. The randomization will be performed by a research assistant with no access to participant information and who did not participate in the enrolment process. The permuted block randomization for a block size of four and six will be used in order to maintain an adequate balance in the number of participants allocated to each of the study groups. The person performing the intervention will be blinded to group allocation. Outcome data will be collected by another two blinded research assistants, one for the intervention group and one for the control group. The completed and coded questionnaires will be entered into databases by research assistant who unaware of group allocation.

The eligible participant will include mothers who have children under 2 years of ages with undernutrition categories residences in Lombok Barat or Lombok Tengah District, mothers who are able to speak Bahasa or Sasak languages, mothers who are able to use a telephone. The exclusion criteria will include mothers with impaired cognitive function, and psychiatric diseases, children suffering from severe/chronic diseases, mental retardation, physical disability, and with hospitalization within six months are excluded from participating in this study.

A priori power analysis has been calculated to determine an adequate sample size for the study. Prior data indicates that the application of the health belief model to teach complementary feeding messages in Ethiopia is 56%. Using a level of conﬁdence of .05 and power of 80% the required sample size was 36.85 participants, with the consideration of 10% dropout rate, it was around 40 for one group. In total the investigator will aim for ﬁnal estimate sample size to be recruited is 80.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have children under 2 years of ages with undernutrition categories residences in Lombok Barat or Lombok Tengah District,
* Mothers who are able to speak Bahasa or Sasak languages,
* Mothers who are able to use a telephone.

Exclusion Criteria:

* Mothers with impaired cognitive function, and psychiatric diseases,
* Children suffering from severe/chronic diseases, mental retardation, physical disability,
* Children with hospitalization within six months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of Undernutrition | before intervention
  The Mother's Knowledge of Child Undernutrition questionnaire. This questionnaire is used to assess mother knowledge related to children undernutrition (Mardani et al., 2014), with Cronbach alpha 0.87. This questionnaire consists of 26 items of questions referring to the definition, types, signs and symptoms, diagnosis, management, and prevention of malnutrition in children. Each question has four answer options (A, B, C, D). A correct answer is scored at one point, while a wrong answer is scored at zero. The sum of answers will be calculated to obtain the total knowledge scores for that participant. The item score ranged from 0 to 26. The higher the score, the greater the understanding related to children's undernutrition
Knowledge of Undernutrition | at two weeks after intervention
  The Mother's Knowledge of Child Undernutrition questionnaire. This questionnaire is used to assess mother knowledge related to children undernutrition (Mardani et al., 2014), with Cronbach alpha 0.87. This questionnaire consists of 26 items of questions referring to the definition, types, signs and symptoms, diagnosis, management, and prevention of malnutrition in children. Each question has four answer options (A, B, C, D). A correct answer is scored at one point, while a wrong answer is scored at zero. The sum of answers will be calculated to obtain the total knowledge scores for that participant. The item score ranged from 0 to 26. The higher the score, the greater the understanding related to children's undernutrition
Complementary Feeding Practice | before intervention
  The complementary feeding practice questionnaire. This questionnaire is used to assess mother's knowledge and competence related to complementary feeding (Hajri et al., 2016), with Cronbach alpha 0.92. This questionnaire contains 29 questions referring to the practice of breastfeeding/complementary feeding, feeding practices based on food safety, responsive feeding practices, and practice of adequate feeding. The answers to this questionnaire are based on two kinds of interval scales: (1) score 0 = if the answer is not recommended, 1 = recommended; and (2) an interval scale with scores of 1 = never, 2 = rarely (1-2 times/week), 3 = sometimes (3-4 times/week), 4 = frequently (5-6 times/week), and 5 = always (every day). The high score indicates that mothers have greater understanding refer to complementary feeding in children. The high score indicates that mothers have greater understanding refer to complementary feeding in children.
Complementary Feeding Practice | at two weeks after intervention
  The complementary feeding practice questionnaire. This questionnaire is used to assess mother's knowledge and competence related to complementary feeding (Hajri et al., 2016), with Cronbach alpha 0.92. This questionnaire contains 29 questions referring to the practice of breastfeeding/complementary feeding, feeding practices based on food safety, responsive feeding practices, and practice of adequate feeding. The answers to this questionnaire are based on two kinds of interval scales: (1) score 0 = if the answer is not recommended, 1 = recommended; and (2) an interval scale with scores of 1 = never, 2 = rarely (1-2 times/week), 3 = sometimes (3-4 times/week), 4 = frequently (5-6 times/week), and 5 = always (every day). The high score indicates that mothers have greater understanding refer to complementary feeding in children. The high score indicates that mothers have greater understanding refer to complementary feeding in children.
Self-efficacy | before intervention
  The self-efficacy questionnaire. This questionnaire is used to assess a mother's self-efficacy in feeding children (Hajri et al., 2016), with Cronbach alpha 0.93. This questionnaire includes 28 questions about a healthy diet and food variety; the amount of food; meal cues; meals based on child development; and general efficacy for feeding children. Each question has scale 0-10. The item score ranged from 0 to 280. The higher the number indicates, the more confident. Research assistants will collect the data before and after the intervention
Self-efficacy | at two weeks after intervention
  The self-efficacy questionnaire. This questionnaire is used to assess a mother's self-efficacy in feeding children (Hajri et al., 2016), with Cronbach alpha 0.93. This questionnaire includes 28 questions about a healthy diet and food variety; the amount of food; meal cues; meals based on child development; and general efficacy for feeding children. Each question has scale 0-10. The item score ranged from 0 to 280. The higher the number indicates, the more confident. Research assistants will collect the data before and after the intervention

SECONDARY OUTCOMES:
Undernutrition (stunting, wasting, and underweight) | before intervention
  Secondary outcomes are undernutrition (stunting, wasting, and underweight). They will be measured using WHO Anthro software version 3.2.2 and expressed as Z-scores for each of the anthropometric indices of undernutrition.
Undernutrition (stunting, wasting, and underweight) | at three months after intervention
  Secondary outcomes are undernutrition (stunting, wasting, and underweight). They will be measured using WHO Anthro software version 3.2.2 and expressed as Z-scores for each of the anthropometric indices of undernutrition.
Undernutrition (stunting, wasting, and underweight) | at six months after intervention
  Secondary outcomes are undernutrition (stunting, wasting, and underweight). They will be measured using WHO Anthro software version 3.2.2 and expressed as Z-scores for each of the anthropometric indices of undernutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, Ph.D, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei County, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol